CLINICAL TRIAL: NCT06237504
Title: The Clinical Efficacy of the Video Laryngeal Mask (SaCoVLM™) in Geriatric Patients: A Comparison With a Conventional Supraglottic Airway Device (Ambu®Auragain™)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1-2023-0081
Record Dates: First submitted 2024-01-22; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Elderly; Laryngeal Mask Airway; General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambu Auragain (Active Comparator): Patients receiving general anesthesia with airway maintained with the 2nd generation SAD, Ambu Auragain.
  Interventions: Device: Ambu®Auragain™
- SaCoVLM (Experimental): Patients receiving general anesthesia with airway maintained with the video LMA, SaCoVLM.
  Interventions: Device: SaCoVLM™

INTERVENTIONS:
Device: SaCoVLM™ — Patients will receive general anesthesia with their airways maintained with the SaCoVLM, which is a newer supraglottic airway device with a video port to directly visualize the upper airway.
  Arms: SaCoVLM
Device: Ambu®Auragain™ — Patients will receive general anesthesia with their airways maintained with the Ambu Auragain, which is a conventional 2nd generation supraglottic airway device.
  Arms: Ambu Auragain

SUMMARY:
This study aims to investigate whether the use of a video LMA device (SacoVLM™) will facilitate successful supraglottic airway device (SAD) insertion compared to the use of a conventional 2nd generation SAD (Ambu®Auragain™) in elderly patients. This study is a randomized trail with a 50% probability of being assigned to either group. Randomization will be done by an anesthesiologist not involved in anesthesia or postoperative outcome assessment. Patients and the investigator in charge of postoperative outcomes assessment will be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

Adult patients 65 years of age or older, ASA class I~III, scheduled for elective surgery under general anesthesia under 2 hours, and eligible for SAD use for airway maintenance.

Exclusion Criteria:

Refusal to participate, patients unable to read consent form, anticipated difficulty in face mask ventilation or airway management based on past history or anatomical structure, upper respiratory tract infection, airway-related diseases such as asthma or pneumonia, risk of gastroesophageal reflux

Min Age: 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Success of SAD insertion on first attempt. | Within the intraoperative period
  The success of SAD insertion is defined as when the a normal square-shaped capnography waveform is detected upon manual ventilation and symmetric movements of the patient's chest wall are observed.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hoon Lee, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No